CLINICAL TRIAL: NCT06464133
Title: Investigation of Filaggrin Gene Mutations Among Latinx Patients With Atopic Dermatitis
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 853590
Record Dates: First submitted 2024-05-10; First posted 2024-06-18 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study, Investigation of Filaggrin Gene Mutations among Latinx patients with Atopic Dermatitis, will examine the association between pathogenic FLG LOF variants and AD in a new population of Latinx patients for which clinical and disease characteristics will be well-described.

DETAILED DESCRIPTION:
Filaggrin deficiency is considered a major target for therapy in Atopic Dermatitis (AD).43 The current status quo with regards to FLG LOF mutations as the strongest known genetic risk factor in AD stems from incomplete data as the majority of studies that have previously examined this association have been carried out in only a limited group of populations (i.e., European ancestry).30 Such partial data impedes our full understanding of genetic risk in AD and consequently has implications for disease prognosis and management. The proposed research represents an attempt to examine long-held paradigms in AD as they relate to genetic risk factors and disease. The development of an independent cohort of Latinx subjects with physician-confirmed diagnosis of AD that is also well phenotyped and grouped by ancestry, while also capturing measures of disease severity, will provide the opportunity to examine a population that has been largely absent from prior studies and further advance our understanding of the pathogenomic role FLG LOF variants in AD.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of AD based on physician report of at least one-year duration
* Self-identification as Latino/Latinx or Hispanic

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who self-identify as Latino/Latinx or Hispanic ethnicity and who have an established diagnosis of AD based on physician report of at least one-year duration will be considered eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify and describe Filaggrin (FLG) loss of function (LOF) variants in the GAD-L cohort using a high-throughput PCR approach that incorporates Fluidigm microfluidics technology and next-generation sequencing (NGS) to sequence the entire FLG gene. | 2 year data/sample collection period - cross-sectional cohort study of patients with a diagnosis of atopic dermatitis

OTHER OUTCOMES:
To examine the correlation between loss of function (LOF) Filaggrin (FLG) mutations and disease onset and severity among Latinx patients with atopic dermatitis (AD). | 2 year data/sample collection period - cross-sectional cohort study of patients with a diagnosis of atopic dermatitis

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No